CLINICAL TRIAL: NCT01785108
Title: Pilot Trial to Preserve Residual Insulin Secretion in Children and Adolescents With Recent Onset Type 1 Diabetes by Using GAD-antigen (Diamyd) Therapy in Combination With Vitamin D and Ibuprofen
Brief Title: DIABGAD - Trial to Preserve Insulin Secretion in Type 1 Diabetes Using GAD-Alum (Diamyd) in Combination With Vitamin D and Ibuprofen
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnny Ludvigsson (Other Government)
Collaborators: Swedish Child Diabetes Foundation (Other); The Research Council of South East Sweden (FORSS) (Unknown); Diamyd Medical AB (Industry)
Responsible Party: Sponsor-Investigator, Johnny Ludvigsson, MD, PhD, Professor, Linkoeping University
Organization: Linkoeping University (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DIABGAD-1
Record Dates: First submitted 2013-02-01; First posted 2013-02-07 (Estimated); Last update posted 2017-08-23 (Actual); Status verified 2017-08

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diamyd; Diabetes; Juvenile Diabetes; Diabetes type 1; Autoimmune Diabetes; Insulin dependent Diabetes; Type 1 diabetes; Type 1 diabetes mellitus; rhGAD65; GAD; GAD65; GAD-alum; Diabetes Mellitus; Diabetes Mellitus, Type 1; Glucose Metabolism Disorders; Metabolic Diseases; Vitamin D; Ibuprofen
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Glucose Metabolism Disorders; Metabolic Diseases | interventions — Vitamin D; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- GAD-Alum (Diamyd) 20µg, Vitamin D and Ibuprofen (Active Comparator): * GAD-Alum (Diamyd) 20 µg given twice with one month interval
  * Vitamin D oral drops, 2000 IU/day, from Day 1 to Day 450
  * Ibuprofen, 400 mg/day, from Day 1 to Day 90
  Interventions: Biological: GAD-Alum (Diamyd) 20 µg; Drug: Vitamin D; Drug: Ibuprofen
- GAD-Alum (Diamyd) 20µg and Vitamin D (Active Comparator): * GAD-Alum (Diamyd) 20 µg given twice with one month interval
  * Vitamin D oral drops, 2000 IU/day, from Day 1 to Day 450
  Interventions: Biological: GAD-Alum (Diamyd) 20 µg; Drug: Vitamin D
- GAD-Alum (Diamyd) 20 µg x 2 and Vitamin D (Active Comparator): * GAD-Alum (Diamyd) 20 µg X 2 given twice with one month interval
  * Vitamin D oral drops, 2000 IU/day, from Day 1 to Day 450
  Interventions: Biological: GAD-Alum (Diamyd) 20 µg X 2; Drug: Vitamin D
- Placebo (Placebo Comparator)
  Interventions: Biological: GAD-Alum (Diamyd) 20 µg X 2; Drug: Vitamin D; Drug: Ibuprofen

INTERVENTIONS:
Biological: GAD-Alum (Diamyd) 20 µg
  Arms: GAD-Alum (Diamyd) 20µg and Vitamin D; GAD-Alum (Diamyd) 20µg, Vitamin D and Ibuprofen
Biological: GAD-Alum (Diamyd) 20 µg X 2
  Arms: GAD-Alum (Diamyd) 20 µg x 2 and Vitamin D; Placebo
Drug: Vitamin D
Drug: Ibuprofen
  Arms: GAD-Alum (Diamyd) 20µg, Vitamin D and Ibuprofen; Placebo

SUMMARY:
The objectives of this study is to

* evaluate the safety and influence of treatment with GAD-Alum (Diamyd) combined with Vitamin D and Ibuprofen on preservation of residual insulin secretion in recently diagnosed Type 1 Diabetes
* evaluate how the above mentioned treatments influence the immune system of the subjects and interact with any viral infections
* evaluate the safety and influence of treatment with double dose of GAD-Alum (Diamyd) plus Vitamin D on the immune system, viral infections, and on preservation of residual insulin secretion in recently diagnosed Type 1 Diabetes

ELIGIBILITY:
Main Inclusion Criteria:

* Male and female patients between 10 and 18 years of age
* Insulin dependent Type 1 Diabetes mellitus diagnosed within the previous 4 months at time of screening
* Fasting C-peptide level at time of screening above or equal to 0.12 nmol/L
* Elevated GAD65 antibodies (GADA) at time of screening

Main Exclusion Criteria:

* Treatment with immunosuppressants, continuous anti-inflammatory drug, Vitamin D or any anti-diabetic medications other than insulin
* A history of certain diseases or conditions (e.g. anemia, HIV, epilepsy, head trauma, neurological diseases or cerebrovascular accident, alcohol or drug abuse etc)
* Treatment with any vaccine within 4 months prior to first planned administration of GAD-Alum/placebo or planned treatment with vaccine up to 4 months after the last injections with GAD-Alum/Placebo, including influenza vaccines
* Participation in other clinical trials with a new chemical entity within the previous 3 months
* Pregnancy or planned pregnancy within 1 year after the last GAD-Alum/placebo dose
* Presence of associated serious disease or condition which in the opinion of the investigator makes the patient non-eligible for the study

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2013-02; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Change in C-peptide (90 minute value and AUC mean 0-120 min) during a Mixed Meal Tolerance Test from baseline to month 6, 15 and 30 | 6 months, 15 months and 30 months

SECONDARY OUTCOMES:
Proportion of patients with a stimulated maximum C-peptide level above 0.2 nmol/L | 6, 15 and 30 months
Hemoglobin A1c (HbA1c), change between baseline and subsequent visits | 6, 15 and 30 months
Exogenous insulin dose per kg body weight and 24 hours, change between baseline and subsequent visits | 6, 15 and 30 months
Th2-deviation of cell-mediated immune response seen, e.g. as increased ratio of IL-5, 10, 13 in comparison with IFN-gamma, TNF-alfa, IL-1 beta, IL-17, and increase of T-regulatory cells | 6, 15 and 30 months
Decrease in inflammatory markers, e.g. TNF-alfa, IL-1 beta, IL-2, IL-17 | 6, 15 and 30 months
Fasting C-peptide, change between baseline and month 6, 15 and 30 | 6, 15 and 30 months

CONTACTS AND LOCATIONS:
Overall Officials: Johnny Ludvigsson, MD,PhD,Prof, Principal Investigator — Linkoeping University
Locations (10):
- Sweden (10):
  - Halmstad Hospital, Halmstad
  - Astrid Lindgren Children's Hospital - Huddinge, Huddinge
  - Kalmar Hospital, Kalmar
  - Linköping University, Linköping
  - Lund University Hospital, Lund
  - Skåne University Hospital, UMAS, Malmo
  - Örebro University Hospital, Örebro
  - Sachsska, Södersjukhuset, Stockholm
  - Astrid Lindgren Children's Hospital, Stockholm
  - Uddevalla Hospital, Uddevalla

REFERENCES:
- [Derived] Ludvigsson J, Routray I, Elluru S, Leanderson P, Larsson HE, Rathsman B, Hanas R, Carlsson A, Ek T, Samuelsson U, Torbjornsdotter T, Aman J, Ortqvist E, Badwal K, Beam C, Casas R. Combined vitamin D, ibuprofen and glutamic acid decarboxylase-alum treatment in recent onset Type I diabetes: lessons from the DIABGAD randomized pilot trial. Future Sci OA. 2020 Jun 23;6(7):FSO604. doi: 10.2144/fsoa-2020-0078. PMID 32802401
- [Derived] Tavira B, Barcenilla H, Wahlberg J, Achenbach P, Ludvigsson J, Casas R. Intralymphatic Glutamic Acid Decarboxylase-Alum Administration Induced Th2-Like-Specific Immunomodulation in Responder Patients: A Pilot Clinical Trial in Type 1 Diabetes. J Diabetes Res. 2018 May 24;2018:9391845. doi: 10.1155/2018/9391845. eCollection 2018. PMID 30009185